CLINICAL TRIAL: NCT06398028
Title: The Preoperative Administration of ICG (Indocyanine Green) Improves Tumor Detection in Patients Undergoing Minimally Invasive Hepatic Resection Guided by Conventional Intraoperative Ultrasound.
Brief Title: The Preoperative Administration of ICG Improves Tumor Detection in Patients Undergoing Minimally Invasive Hepatic Resection Guided by Conventional Intraoperative Ultrasound.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LIVERGREEN
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Liver Tumor; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Multicentric low-intervention phase IV clinical trial of preoperative ICG administration for intraoperative detection of liver tumors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green has a sharply defined spectral peak absorption of near-infrared light at 800 nm in blood plasma or blood. This is the same wavelength at which the optical density of oxygenated hemoglobin in blood approximately equals that of reduced hemoglobin. Therefore, this coincidental light absorption makes it possible to measure indocyanine green concentrations in blood, plasma and serum in terms of its optical density at 800 nm, independent of variations in oxygen saturation level

SUMMARY:
Summary:

Preoperative administration of indocyanine green (ICG) improves the detection of liver tumors in patients undergoing minimally invasive liver resection guided by conventional intraoperative ultrasound. The primary objectives of this study are to evaluate the efficacy of ICG fluorescence uptake in combination with intraoperative ultrasonography and preoperative magnetic resonance imaging for detecting liver tumors. Additionally, a machine-learning algorithm will be developed to enhance liver tumor detection using ICG through photographic analysis. Secondary objectives include investigating the distribution of ICG in liver tissue and its correlation with hepatic fibrosis and steatosis, as well as describing patterns of ICG uptake and their relationship with liver tumors. The study also aims to analyze various clinical outcomes such as the 30-day comprehensive complication index, operation time, conversion to open surgery rate, length of hospital stay, liver tumor recurrence, readmission rate, complications, and 90-day mortality. This research seeks to advance tumor detection methods and improve patient outcomes in minimally invasive liver resection procedures.

ELIGIBILITY:
Inclusion Criteria

* Patients with liver tumors with an indication for minimally invasive surgery, evaluated by the hospital's multidisciplinary liver tumor board (MDTB).
* Contrast enhanced MRI within 6 weeks prior to liver surgery
* ≥18 years old
* Absence of exclusion criteria and able to provide consent for data collection and analysis

Exclusion Criteria

* Emergency surgery
* Patients in which ICG is contraindicated: previous history of iodine hypersensitivity, patients with renal failure (GFR <60 mL/min/1.73 m2), uremia, clinical hyperthyroidism, autonomic thyroid adenomas, or focal and diffuse autonomic abnormalities of the thyroid gland.
* Previous liver surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
Number of liver tumors identified intraoperatively using preoperative magnetic resonance imaging, intraoperative ultrasound, and ICG fluorescence. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes